CLINICAL TRIAL: NCT02205086
Title: Empowering Physicians With Evidence-Based Decision Support for Pediatric Rheumatology
Acronym: Rheumatology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SimulConsult, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SimulConsult2
Record Dates: First submitted 2014-07-25; First posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnosis (Other): Test diagnostic decision support software
  Interventions: Other: Diagnosis

INTERVENTIONS:
Other: Diagnosis — Unaided: The testers will record a differential diagnosis consisting of a list of diseases and their ranking and a prioritized list of test orders, as well as the most appropriate referral for further evaluation and treatment of the patient.
  Aided: Then testers will enter the case into diagnostic decision support software and after getting advice from the software, the testers will record the same information as in Unaided, but allowing for the possibility that responses could differ as a result of using the software.

SUMMARY:
This study compares the ability of clinicians to make diagnoses with or without the assistance of diagnostic decision support software. The area of clinical focus is primarily rheumatology.

DETAILED DESCRIPTION:
The study uses written case vignettes, not decisions about patients seeking care from the study subjects (i.e., clinicians).

ELIGIBILITY:
Inclusion criteria: Clinicians in various medical specialties

Exclusion criteria: Non-clinician

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Measures of Diagnostic effectiveness | Completion of each case vignette (typically ½ hour)
  Each clinician subject reviews each case vignette and lists their differential diagnosis ("Unaided").
  Then the clinician subject uses the diagnostic decision support software and then lists a revised differential diagnosis ("Aided").
  The match between the clinician subject's differential diagnosis and a Gold Standard differential diagnosis list for each case is measured, looking at rank order of correct diseases and omissions.

SECONDARY OUTCOMES:
Measures of Patient workup effectiveness | Completion of each case vignette (typically in the same ½ hour as measure 1)
  Each clinician subject reviews each case vignette and lists their initial workup ("Unaided").
  Then the clinician subject uses the diagnostic decision support software and then lists a revised initial workup ("Aided").
  The match between the clinician subject's initial workup and a Gold Standard workup list for each case is measured, looking at rank order of correct diseases and omissions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Segal, MD PhD, Principal Investigator — SimulConsult, Inc.
Locations (1):
- SimulConsult, Brookline, Massachusetts, United States

REFERENCES:
- [Background] Segal MM, Williams MS, Gropman AL, Torres AR, Forsyth R, Connolly AM, El-Hattab AW, Perlman SJ, Samanta D, Parikh S, Pavlakis SG, Feldman LK, Betensky RA, Gospe SM Jr. Evidence-based decision support for neurological diagnosis reduces errors and unnecessary workup. J Child Neurol. 2014 Apr;29(4):487-92. doi: 10.1177/0883073813483365. Epub 2013 Apr 10. PMID 23576414
- [Background] Segal MM, Schiffmann R. Decision support for diagnosis: co-evolution of tools and resources. Neurology. 2012 May 15;78(20):1546-7. doi: 10.1212/WNL.0b013e3182563c36. Epub 2012 Apr 18. No abstract available. PMID 22517101
- [Derived] Segal MM, Athreya B, Son MB, Tirosh I, Hausmann JS, Ang EY, Zurakowski D, Feldman LK, Sundel RP. Evidence-based decision support for pediatric rheumatology reduces diagnostic errors. Pediatr Rheumatol Online J. 2016 Dec 13;14(1):67. doi: 10.1186/s12969-016-0127-z. PMID 27964737